CLINICAL TRIAL: NCT02280720
Title: A Randomized Prospective Multicenter Trial to Compare Vascular Healing and Vasodilation at 2 Months After Deployment of TItanium-nitride-oxide-coated OPTIMAX™ Stent and PROMUS-ELEMENT™ Drug-Eluting Stent in Patients With Acute Coronary Syndromes by Means of Optical Coherence Tomography and Coronary Flow Reserve
Brief Title: Vascular Healing After Deployment of Titanium-nitride-oxide-coated OPTIMAX™ Stent and PROMUS-ELEMENT™ Everolimus-Eluting Stent
Acronym: TIDES-OCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital District of Satakunta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SA-006
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Acute Coronary Syndrome
Keywords: titanium-nitride-oxide-coated stent; everolimus-eluting stent; optical coherence tomography; strut coverage
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CoCr-BAS (Active Comparator): Stenting using Optimax™ cobalt-chromium alloy platform with a titanium-nitride-oxide coating
  Interventions: Procedure: Stenting using Optimax™
- PtCr-EES (Active Comparator): Stenting using PROMUS Element™ Plus durable polymer everolimus-eluting stent built on a platinum-chromium platform.
  Interventions: Procedure: Stenting using PROMUS Element™ Plus

INTERVENTIONS:
Procedure: Stenting using Optimax™
  Arms: CoCr-BAS
Procedure: Stenting using PROMUS Element™ Plus
  Arms: PtCr-EES

SUMMARY:
The purpose of this study is to compare vascular healing of the stented segment after deployment of titanium-nitride-oxide coated cobalt-chromium Optimax™-stent stent and Promus-Element™ everolimus-eluting stent in patients with acute coronary syndromes requiring percutaneous coronary intervention.

1. Comparison of OCT and CFR findings of titanium-nitride-oxide coated cobalt-chromium Optimax™-stent and Promus-Element™ everolimus-eluting stent at two months after the index procedure.
2. Comparison of intravascular coronary flow reserve measurement to non-invasive transthoracic echocardiography-derived coronary flow reserve measurement.
3. Comparison of epicardial vasodilation to coronary microcirculatory vasodilation

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and <80 years
2. STEMI or NSTEMI (assumed by investigator to be type 1 myocardial infarction, according to universal definitions of MI; EHJ 2007; 28(20):2525-38); or unstable angina (clinical symptoms of chest pain, ecg suggestive of reversible ischemia)
3. Patient is willing to comply with specified follow-up evaluations
4. Patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent, approved by the appropriate Medical Ethics committee or Institutional Review Board
5. Single de novo or non-stented restenosis lesion
6. Patients with two-vessel disease may have undergone successful treatment of the non-target vessel with approved devices up to and including the index procedure but must be prior to the index target vessel treatment
7. Target lesion (maximum 20 mm length by visual estimation) to be covered by a single stent of maximum 23mm length
8. Reference vessel diameter must be >2.5mm and <4.0mm by visual estimate.
9. The vessel diameter should be measured after pre-dilation procedure and after intracoronary nitroglycerin if vasospasm is suspected
10. Target lesion >50% and <100% stenosed by visual estimate

Exclusion Criteria:

1. Pre-existing diagnosis of diabetes irrespective of its type
2. Impaired renal function (serum creatinine >177micromol/l) or on dialysis
3. Platelet count < 10 e5 cells/mm3
4. Patient has a history of bleeding diathesis or coagulopathy or patients in whom antiplatelet and and/or anticoagulation therapy is contraindicated
5. Patient has received organ transplant or is on a waiting list for any organ transplant
6. Patient has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/prasugrel, stainless steel alloy, or contrast agent that cannot be adequately pre-medicated
7. Patient presents with cardiogenic shock
8. Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study
9. Currently participating in another intestigational drug or device study
10. Unprotected left main disease
11. Ostial target lesions
12. Chronic total occlusion
13. Calcified target lesions that cannot be adequately pre-dilated
14. Target lesion has excessive tortuosity unsuitable for stent delivery and deployment
15. Target lesion involving bifurcation with a side branch larger than 2.0mm in diameter
16. A >30% stenosis proximal or distal to the target lesion that cannot be covered with the same stent
17. Diffuse distal disease
18. Prior stent in the target vessel

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of uncovered struts | 2 months

SECONDARY OUTCOMES:
Coronary flow reserve | 2 months

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (4):
  - Kokkola Central Hospital, Kokkola
  - Heart Center, Kuopio University Hospital, Kuopio
  - Heart Center, Satakunta Central Hospital, Pori
  - Heart Center, Turku University Hospital, Turku